CLINICAL TRIAL: NCT07028528
Title: A Randomized Placebo Controlled Trial Assessing the Efficacy of Levagen+ for Treating Symptoms of Diabetic Peripheral Neuropathy
Brief Title: Levagen+ Efficacy Study on Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Gencor Pacific Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEULEV
Record Dates: First submitted 2025-05-15; First posted 2025-06-19 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — palmidrol

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, placebo-controlled, parallel dose response study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levagen+ (Experimental): Take 1 capsule twice daily with water after food. Each capsule will contain:
  A175mg containing 150 mg of palmitoylethanolamide (PEA). Total daily dose of 350mg Levagen+ containing 300 mg PEA.
  Interventions: Dietary Supplement: Levagen+
- Placebo (Placebo Comparator): Take 1 capsule twice daily with water after food. Each capsule will contain microcrystalline cellulose [MCC].
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Levagen+ — Participants will take 1 capsule twice daily with water after food. Each capsule will contain: A175mg containing 150 mg of palmitoylethanolamide (PEA). Total daily dose of 350mg Levagen+ containing 300 mg PEA
  Other Names: palmitoylethanolamide; PEA
  Arms: Levagen+
Other: Placebo — Participants will take 1 capsule twice daily with water after food. Each capsule will contain microcrystalline cellulose [MCC]
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the efficacy of Levagen+ supplementation for the symptoms of diabetic peripheral neuropathy (DPN) in patients with DPN.

Participants will have remote visits and attend a local pathology centre for blood draws. They will take the study product for 12 weeks, from baseline to week 12 they will have remote visits every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years.
* Using prescribed glucose-lowering medications, including oral medications (stable dose for 3 months or more) and/or insulin for diabetes (type 1 or 2).
* Scoring12 or more on the Self-reported Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS).
* Able to provide informed consent.
* Agree not to change current diet and/or exercise frequency or intensity during entire enrolment period.
* Agree to not participate in another clinical trial during the study period.
* Able to attend an ACL collection centre.

Exclusion Criteria:

* Peripheral neuropathy due to causes other than diabetes mellitus (e.g. nutritional deficiencies; hereditary sensory neuropathy; paraneoplastic diseases; advanced liver disease; kidney disease; hypothyroidism; prolonged phenytoin, warfarin or immunosuppressive drug use; active infection [HIV, Lyme disease, Epstein-Barr virus, Hepatitis C, Shingles, Leprosy]; autoimmune disease [Sjogren syndrome, Lupus, Rheumatoid arthritis, Guillain-Barre syndrome]; trauma / injury; toxins [heavy metals, chemicals]; antibiotics; or inflammatory conditions [vasculitis]).
* Serious illness e.g., paraneoplastic diseases, advanced liver disease, kidney disease, hypothyroidism, mood disorders such as depression, anxiety or bipolar disorder, neurological disorders such as MS, or heart conditions, or peripheral vascular disease
* Unstable illness e.g., diabetes and thyroid gland dysfunction, hypercholesterolemia
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years.
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy including low dose aspirin
* Herbal medicines for pain relief including, but not limited to, medicinal cannabis, willow bark (Salix alba), Boswellia (Boswellia serrata) or turmeric/curcumin (Curcuma longa).
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse.
* Chronic past and/or current alcohol use (>14 alcoholic drinks per week)
* Females attempting to conceive, pregnant or lactating
* Allergic, sensitive or intolerant to any of the ingredients in active or placebo formula.
* Difficulty swallowing capsules.
* Participants who are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 1 month.
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the end of the study period in overall severity of neuropathic pain | Baseline to week 12
  Change from baseline to the end of the study period in overall severity of neuropathic pain, as assessed by the Brief Pain Inventory Short Form for Diabetic Peripheral Neuropathy (BPI-DPN).
  This is a self-reported scale, higher scores indicate greater pain and interference.

SECONDARY OUTCOMES:
Change from baseline to the end of the study period in Neuropathic Pain Symptom Inventory | Baseline to week 12
  Change from baseline to the end of the study period in Neuropathic Pain Symptom Inventory (NPSI). This is a self-administered questionnaire used to evaluate neuropathic pain intensity across 5 categories, namely "superficial spontaneous pain", "deep spontaneous pain", "paroxysmal pain", "evoked pain", and "dysesthesia / paraesthesia". There are 10 pain descriptors and 2 items related to abnormal sensations. The scale ranges from 0 (no pain at all) to 10 (worst pain imaginable). The total scores of all items are combined to find the total pain intensity
Change from baseline to the end of the study period in Safety via Adverse Event reporting | Baseline to week 12
  Change from baseline to the end of the study period in safety via Adverse Event reporting and incident rate ratio between placebo and Levagen+
Change from baseline to the end of the study period in Safety Markers (FBC) | Baseline to week 12
  Change from baseline to the end of the study period in safety Markers (FBC - Full Blood Count) via blood test.
Change from baseline to the end of the study period in Safety Markers (E/LFT) | Baseline to week 12
  Change from baseline to the end of the study period in safety Markers (E/LFT) via blood test.
Change from baseline to the end of the study period in Safety (Vitals - BP) | Baseline to week 12
  Change from baseline to the end of the study period in Safety Markers vital signs (blood pressure)
Change from baseline to the end of the study period in Safety (Vitals - heart rate) | Baseline to week 12
  Change from baseline to the end of the study period in Safety Markers vital signs (heart rate)
Change from baseline to the end of the study period in Medical Outcomes Study - Sleep Scale (MOS-Sleep) | Baseline to week 12
  Change from baseline to the end of the study period in Medical Outcomes Study - Sleep Scale (MOS-Sleep). This is a self-administered 12-item questionnaire that includes a Sleep Problem Index and evaluates 6 dimensions of sleep difficulty, namely: "sleep disturbance", "sleep adequacy", somnolence", "quantity of sleep/optimal sleep", "awakening short of breath or with headache", and "occurrence of snoring". The Sleep Problem Index summarises information across 9 items and is rated on a scale of 1 (all of the time) to 6 (none of the time).
Change from baseline to the end of the study period in Depression Anxiety and Stress Scale (DASS-21) | Baseline to week 12
  Change from baseline to the end of the study period in Depression Anxiety and Stress Scale (DASS-21). The DASS-21 is a self-reported questionnaire derived from the original 42-item DASS and is a quantitative measure of distress. It consists of 3 subscales: the depression subscale (DASS-D), anxiety subscale (DASS-A) and stress subscale (DASS-S). Each subscale contains 7 items which are rated on a 4-point severity/frequency scale. The scores for each subscale are calculated by summing the scores for the relevant items. Higher scores indicate greater distress.
Change from baseline to the end of the study period in Glycaemic control (HbA1c) | Baseline to week 12
  Change from baseline to the end of the study period in Glycaemic control (HbA1c)
Change from baseline to the end of the study period in Glycaemic control (fasting blood glucose) | Baseline to week 12
  Change from baseline to the end of the study period in Glycaemic control (fasting blood glucose)
Change from baseline to the end of the study period in Anthropometry (weight) | Baseline to week 12
  Change from baseline to the end of the study period in Anthropometry (weight).
Change from baseline to the end of the study period in Anthropometry (height) | Baseline to week 12
  Change from baseline to the end of the study period in Anthropometry (height).
Change from baseline to the end of the study period in Anthropometry (BMI) | Baseline to week 12
  Change from baseline to the end of the study period in Anthropometry (BMI).
Change from baseline to the end of the study period in use of rescue medication for pain | Baseline to week 12
  Change from baseline to the end of the study period in use of rescue medication for pain. Participants will be allowed to use a rescue medication as needed, with use documented via participant diaries including date, time, dosage, reason for use. Data will be analysed based on total usage, frequency, and the proportion of participants requiring rescue medication.

CONTACTS AND LOCATIONS:
Overall Officials: Ramasamy Venkatesh, Study Director — Gencor Pacific
Locations (1):
- RDC Clinical, Fortitude Valley, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided